CLINICAL TRIAL: NCT02035696
Title: A Phase I/II, Randomized, Observer-Blind, Multicenter Study to Evaluate Immunogenicity and Safety of Four Influenza Vaccines in Healthy Pediatric Subjects 6 to < 48 Months of Age.
Brief Title: Safety and Immunogenicity of a Four Influenza Vaccines in Children Ages 6 Months Old to Less Than 48 Months Old
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V58P16; 2013-002081-39 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-14 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: influenza; children; safety; tolerability; immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TIVc-High Dose (Experimental): Subjects (6 to <48 months old) received two doses of 0.75 mL of TIVc vaccine
  Interventions: Biological: Trivalent influenza vaccine (TIVc)
- TIVc-Full Dose (Experimental): Subjects(6 to <48 months old) received two doses of 0.50 mL of TIVc vaccine
  Interventions: Biological: Trivalent influenza vaccine (TIVc)
- TIVc- Half Dose (Experimental): Subjects (6 to <48 months old)received two doses of 0.25 mL of TIVc vaccine
  Interventions: Biological: Trivalent influenza vaccine (TIVc)
- TIVe (Active Comparator): Subjects (6 to <48 months old) received two doses of TIVe vaccine(IM/0.25mL -for ages 6 to <36 months and IM/ 0.5 mL -for ages 36 to <48 months)
  Interventions: Biological: Trivalent influenza vaccine-licensed

INTERVENTIONS:
Biological: Trivalent influenza vaccine (TIVc)
  Arms: TIVc- Half Dose; TIVc-Full Dose; TIVc-High Dose
Biological: Trivalent influenza vaccine-licensed — Licensed influenza vaccine
  Arms: TIVe

SUMMARY:
To evaluate the safety and immunogenicity of four influenza vaccines in children 6 months to < 48 months of age

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject, male or female, 6 through < 48 months of age at the time of enrollment, who has never previously received an influenza vaccine
* Individual who has a parent or guardian that can give written informed consent after understanding the nature of the study and are available for follow-up

Exclusion Criteria:

* Individuals recently vaccinated against influenza
* Subjects with contraindications to receive influenza vaccine

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 671 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (21):
  - Site 116, Phoenix, Arizona
  - Site 119, Tucson, Arizona
  - Site 109, Little Rock, Arkansas
  - Site 112, Long Beach, California
  - Site 113, Ontario, California
  - Site 117, San Diego, California
  - Site 114, West Covina, California
  - Site 107, Thornton, Colorado
  - Site 111, Miami, Florida
  - Site 108, Miami Beach, Florida
  - Site 121, Gainesville, Georgia
  - Site 101, Omaha, Nebraska
  - Site 104, Omaha, Nebraska
  - Site 105, Omaha, Nebraska
  - Site 106, Omaha, Nebraska
  - Site 103, Youngstown, Ohio
  - Site 102, Charleston, South Carolina
  - Site 115, Houston, Texas
  - Site 110, Salt Lake City, Utah
  - Site 118, St. George, Utah
  - Site 120, Spokane, Washington
- Finland (2):
  - Site 502, Kuopio
  - Site 506, Tampere
- Philippines (2):
  - Site 302, City of Muntinlupa
  - Site 301, Manila
- Thailand (2):
  - Site 201, Bangkok
  - Site 202, Bangkok

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 centers in the United States, 1 center in Finland, 2 centers in Thailand, 2 centers in Philippines
Pre-assignment Details: All enrolled Subjects were included in the trial
Groups:
- TIVe: Subjects (6 to <48 months old) received two doses of TIVe vaccine
Period: Overall Study
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Started | 174 | 166 | 167 | 164
Completed | 171 | 163 | 164 | 161
Not Completed | 3 | 3 | 3 | 3
Not completed — Lost to Follow-up | 0 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe | Total
Number analyzed (Participants) | 174 | 166 | 167 | 164 | 671
Age, Continuous [Mean (Standard Deviation); unit: Months] | 25.3 (11.5) | 25.0 (11.5) | 25.6 (11.5) | 25.3 (11.9) | 25.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 84 | 82 | 77 | 87 | 330
  MALE | 90 | 84 | 90 | 77 | 341

OUTCOME MEASURES:

1. Primary Outcome: Ratios of Geometric Mean Titer (GMT) in Subjects (6 to <48 Months Old) After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of ratios of GMTs in subjects (6 to <48 months old), measured by hemagglutination inhibition (HI) assay, day 1 to day 50 after vaccination with two doses of either TIVc or TIVe vaccine
Time Frame: Day 50/Day 1
Population: Analysis was done on Per Protocol (PP) population i.e. all subjects in the FAS Efficacy/Immunogenicity Set who are not excluded due to reasons defined prior to unblinding or analysis
Measure: Number (95% Confidence Interval); unit: Ratios
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 156 | 147 | 141 | 145
Ratios
  A/H1N1 | 7.82 [4.3 to 14.21] | 5.5 [3.01 to 10.04] | 5.93 [3.21 to 10.96] | 3.69 [2.02 to 6.74]
  A/H3N2 | 10.53 [6.34 to 17.49] | 10.84 [6.5 to 18.07] | 6.47 [3.84 to 10.9] | 11.95 [7.17 to 19.91]
  B | 5.18 [3.73 to 7.96] | 4.27 [2.77 to 6.58] | 3.87 [2.49 to 6.02] | 6.65 [4.32 to 10.25]
Statistical Analysis 1: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of a TIVc-High Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H1N1 at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 0.99, 95% CI 2-sided [0.65 to 1.52]
Statistical Analysis 2: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of a TIVc-High Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H1N1 at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group ratios at Day 50 = 2.11, 95% CI 2-sided [1.5 to 2.98]
Statistical Analysis 3: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of a TIVc-High Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H3N2 at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group ratios at Day 1 = 0.68, 95% CI 2-sided [0.43 to 1.06]
Statistical Analysis 4: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of a TIVc-High Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H3N2 at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 50 = 0.71, 95% CI 2-sided [0.58 to 0.87]
Statistical Analysis 5: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of a TIVc-High Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain B at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 1, 95% CI 2-sided [0.92 to 1.08]
Statistical Analysis 6: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of a TIVc-High Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain B at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group ratios at Day 50 = 0.78, 95% CI 2-sided [0.6 to 1.01]
Statistical Analysis 7: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of a TIVc-Full Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H1N1 at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 1.27, 95% CI 2-sided [0.83 to 1.96]
Statistical Analysis 8: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of a TIVc-Full Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H1N1 at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 50 = 1.6, 95% CI 2-sided [1.13 to 2.28]
Statistical Analysis 9: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of a TIVc-Full Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H3N2 at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 0.52, 95% CI 2-sided [0.33 to 0.81]
Statistical Analysis 10: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of a TIVc-Full Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H3N2 at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 50 = 0.64, 95% CI 2-sided [0.52 to 0.78]
Statistical Analysis 11: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of a TIVc-Full Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain B at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group ratios at Day 1 = 0.96, 95% CI 2-sided [0.89 to 1.04]
Statistical Analysis 12: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of a TIVc-Full Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain B at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 50 = 0.64, 95% CI 2-sided [0.49 to 0.84]
Statistical Analysis 13: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of a TIVc- Half Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H1N1 at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 1.02, 95% CI 2-sided [0.66 to 1.58]
Statistical Analysis 14: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of a TIVc- Half Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H1N1 at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group ratios at Day 50 = 1.62, 95% CI 2-sided [1.14 to 2.3]
Statistical Analysis 15: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of a TIVc- Half Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H3N2 at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 0.74, 95% CI 2-sided [0.47 to 1.17]
Statistical Analysis 16: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of a TIVc- Half Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain A/H3N2 at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group ratios at Day 50 = 0.46, 95% CI 2-sided [0.38 to 0.57]
Statistical Analysis 17: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of a TIVc- Half Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain B at Day 1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 1 = 0.94, 95% CI 2-sided [0.87 to 1.02]
Statistical Analysis 18: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of a TIVc- Half Dose to TIVe, assessed in terms of vaccine group GMT ratios against influenza strain B at Day 50; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI of the vaccine group GMT ratio ≥ 0.67; Vaccine Group Ratios at Day 50 = 0.57, 95% CI 2-sided [0.44 to 0.75]

2. Primary Outcome: Percentages of Subjects (6 to <48 Months Old) Achieving Seroconversion or Significant Increase After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms number (%) of subjects (6 to <48 months old) achieving seroconversion as measured by HI antibody titer, day 50 after vaccination with two doses of either TIVc or TIVe vaccine Seroconversion was defined as subjects with either a pre-vaccination (baseline) HI titer < 1:10 and post-vaccination HI titer ≥ 1:40 or with a pre-vaccination HI titer ≥ 1:10 and a ≥ 4-fold increase in post-vaccination HI antibody titer
Time Frame: Day 50 post vaccination
Population: Analysis was done on PP population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 156 | 147 | 141 | 145
Percentages of subjects
  A/H1N1_Day 50 | 83 [77 to 89] | 81 [74 to 87] | 79 [72 to 86] | 74 [66 to 81]
  A/H3N2_Day 50 | 94 [89 to 97] | 90 [84 to 94] | 87 [80 to 92] | 92 [87 to 96]
  B_Day 50 | 69 [61 to 76] | 69 [61 to 77] | 62 [54 to 70] | 80 [73 to 86]
Statistical Analysis 1: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of TIVc-High Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain A/H1N1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the Lower limit of the 2-sided 95% CI on the difference between seroconversion rates ≥ -10%; Vaccine Group Differences = 10, 95% CI 2-sided [0 to 18.9]
Statistical Analysis 2: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of TIVc-High Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain A/H3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group Differences = 2, 95% CI 2-sided [-4 to 8]
Statistical Analysis 3: Comparison: TIVc-High Dose vs TIVe; Non-inferiority of immune responses of TIVc-High Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group differences = -11, 95% CI 2-sided [-21.1 to -1.5]
Statistical Analysis 4: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of TIVc-Full Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain A/H1N1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group Differences = 7, 95% CI 2-sided [-2.5 to 16.8]
Statistical Analysis 5: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of TIVc-Full Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain A/H3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group differences = -3, 95% CI 2-sided [-9.5 to 4.1]
Statistical Analysis 6: Comparison: TIVc-Full Dose vs TIVe; Non-inferiority of immune responses of TIVc-Full Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group Differences = -11, 95% CI 2-sided [-20.5 to -1]
Statistical Analysis 7: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of TIVc- Half Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain A/H1N1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group Differences = 6, 95% CI 2-sided [-4.2 to 15.4]
Statistical Analysis 8: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of TIVc- Half Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain A/H3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group Differences = -6, 95% CI 2-sided [-13.4 to 1.3]
Statistical Analysis 9: Comparison: TIVc- Half Dose vs TIVe; Non-inferiority of immune responses of TIVc- Half Dose to TIVe, assessed in terms of Vaccine Group Differences with seroconversion against influenza strain B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Vaccine Group Differences = -18, 95% CI 2-sided [-27.8 to -7.2]

3. Primary Outcome: Desirability Index Score of Subjects (6 to <48 Months Old) Reporting Severe Solicited Local and Systemic Reactions After Vaccination With Either TIVc or TIVe Vaccine
Description: Differences in percentages of subjects (6 to <48 months old) with severe local solicited AEs and severe solicited systemic AEs, 3 days after vaccination with either TIVc or TIVe vaccine was assessed in terms of an individual desirability index score (High dose, Full dose, Half dose TIVc vs. TIVe vaccine). An individual desirability index score was assigned to each (non-transformed) safety value based on predefined functions. Each desirability index score is assigned a value between 0 and 1, wherein 0 is an undesirable response and 1 is a highly desirable response.
Time Frame: Day 1 to Day 3
Population: Analysis was done on PPSd-All subjects in the FASd who:Correctly received the vaccine (i.e., received the vaccine to which the subjects is randomized and at the scheduled time points).
Measure: Number; unit: percentage of participants
Groups:
- TIVc-High Dose-TIVe: Subjects (6 to <48 months old) received two doses of 0.75 mL of TIVc vaccine vs Subjects (6 to <48 months old) received two doses of TIVe vaccine
- TIVc-Full Dose-TIVe: Subjects(6 to <48 months old) received two doses of 0.50 mL of TIVc vaccine vs Subjects (6 to <48 months old) received two doses of TIVe vaccine
- TIVc- Half Dose-TIVe: Subjects (6 to <48 months old)received two doses of 0.25 mL of TIVc vaccine vs Subjects (6 to <48 months old) received two doses of TIVe vaccine
Arm/Group | TIVc-High Dose-TIVe | TIVc-Full Dose-TIVe | TIVc- Half Dose-TIVe
Number analyzed (Participants) | 305 | 294 | 291
percentage of participants
  Severe solicited local AEs | 0.000 | 0.000 | 0.000
  Severe solicited systemic AEs | 0.040 | 0.000 | 0.000
Statistical Analysis 1: Comparison: TIVc-High Dose-TIVe; Test type: Superiority or Other; Desirability Index Score = 0.000 — Desirability Score: If this difference is negative, then it is defined as non-desirable (D equal to 0), while if the difference is positive, then D will equal to the relative reduction calculated in the following way: D = (TIVe - TIVc Dose )/TIVe
Statistical Analysis 2: Comparison: TIVc-Full Dose-TIVe; Test type: Superiority or Other; Desirability Index Score = 0.000 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: TIVc- Half Dose-TIVe; Test type: Superiority or Other; Desirability Index Score = 0.000 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percentages of Subjects (6 to <48 Months Old) Achieving Seroconversion or Significant Increase After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of number (%) of subjects (6 to <48 months old) achieving seroconversion as measured by HI assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
  Seroconversion was defined as subjects with either a pre-vaccination (baseline) HI titer < 1:10 and post-vaccination HI titer ≥ 1:40 or with a pre-vaccination HI titer ≥ 1:10 and a ≥ 4-fold increase in post-vaccination HI antibody titer
  The Center for Biologics Evaluation, Research, and Review (CBER) criterion for pediatric population is that the lower bound of the two-sided 95% confidence interval (CI) for the percentage of subjects achieving seroconversion for HI antibody should meet or exceed 40%
  The Committee for Medicinal Products for Human Use (CHMP) criterion for pediatric population is that the percentage of subjects achieving seroconversion or significant increase in HI antibody titers >40%
Time Frame: Day 50 post vaccination
Population: Analysis was done on Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 170 | 164 | 161 | 159
Percentages of subjects
  A/H1N1 | 84 [77 to 89] | 80 [74 to 86] | 82 [75 to 88] | 73 [65 to 80]
  A/H3N2 | 94 [89 to 97] | 91 [85 to 95] | 88 [81 to 92] | 93 [88 to 96]
  B | 68 [61 to 75] | 70 [62 to 76] | 63 [55 to 70] | 79 [72 to 85]

5. Secondary Outcome: Percentages of Subjects (6 to <48 Months Old) Achieving HI Titer ≥1:40 After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of number (%) of subjects (6 to <48 months old) achieving HI titer ≥1:40 as measured by HI assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
  The CBER criterion for pediatric population is that the lower bound of the two-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 70%
  The CHMP criterion for pediatric population is that the percentage of subjects achieving HI antibody titers ≥1:40 should be >70%
Time Frame: Day 1, Day 50 post vaccination
Population: Analysis was done on FAS
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 170 | 164 | 161 | 159
Percentages of subjects
  A/H1N1: Day 1 | 26 [20 to 34] | 32 [25 to 39] | 29 [22 to 37] | 26 [20 to 34]
  A/H1N1: Day 50 | 86 [80 to 91] | 85 [78 to 90] | 86 [79 to 91] | 77 [69 to 83]
  A/H3N2: Day 1 | 45 [37 to 53] | 40 [33 to 48] | 48 [41 to 56] | 52 [44 to 60]
  A/H3N2: Day 50 | 98 [95 to 100] | 98 [94 to 99] | 97 [93 to 99] | 99 [97 to 100]
  B: Day 1 | 2 [0 to 5] | 0 [0 to 2] | 1 [0.016 to 3] | 3 [1 to 7]
  B: Day 50 | 69 [61 to 76] | 70 [62 to 76] | 63 [55 to 70] | 80 [73 to 86]

6. Secondary Outcome: Geometric Mean Ratios (GMR) in Subjects (6 to <48 Months Old) After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of GMR in subjects (6 to <48 months old) as measured by HI assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
  The CHMP criterion is mean geometric ratio (GMR) >2.5
Time Frame: Day 50 post vaccination over day 1
Population: Analysis was done on FAS
Measure: Number (95% Confidence Interval); unit: Ratios
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 170 | 164 | 161 | 159
Ratios
  A/H1N1 | 12 [7.05 to 19] | 8.58 [5.08 to 14] | 8.94 [5.28 to 15] | 5.14 [3.04 to 8.68]
  A/H3N2 | 12 [7.83 to 19] | 13 [8.05 to 20] | 7.68 [4.91 to 12] | 14 [8.83 to 22]
  B | 6.14 [4.27 to 8.84] | 5.29 [3.64 to 7.7] | 4.72 [3.24 to 6.88] | 7.57 [5.21 to 11]

7. Secondary Outcome: Geometric Mean Ratios (GMR) in Subjects (6 to <48 Months Old) After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of GMR in subjects (6 to <48 months old) as measured by MN assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
Time Frame: Day 50 post vaccination over day 1
Population: Analysis was done on PPS
Measure: Number (95% Confidence Interval); unit: Ratios
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 156 | 148 | 141 | 147
Ratios
  A/H1N1 | 7.84 [4.29 to 14.33] | 5.81 [3.17 to 10.65] | 5.98 [3.22 to 11.09] | 17.82 [9.73 to 32.62]
  A/H3N2 | 8.4 [5 to 14.12] | 8.97 [5.32 to 15.12] | 5.58 [3.28 to 9.51] | 8.9 [5.28 to 14.98]
  B | 12.78 [8.09 to 20.2] | 10.43 [6.58 to 16.52] | 9.99 [6.25 to 15.99] | 17.55 [11.08 to 27.78]

8. Secondary Outcome: Percentages of Subjects (6 to <48 Months Old) With High Post Vaccination HI Titers (i.e. HI Titers ≥1:110, ≥1:150, ≥1:330 and ≥1:629) After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of number (%) of subjects (6 to <48 months old) achieving post vaccination HI titers (i.e. HI titers ≥1:110, ≥1:150, ≥1:330 and ≥1:629) as measured by HI assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
Time Frame: Day 1 and Day 50 post vaccination
Population: Analysis was done on PPS
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 156 | 147 | 141 | 145
Percentages of subjects
  A/H1N1: Day 1: HI titers ≥1:110 | 26 [19 to 33] | 31 [24 to 39] | 26 [19 to 34] | 26 [19 to 33]
  A/H1N1: Day 50: HI titers ≥1:110 | 78 [70 to 84] | 80 [72 to 86] | 71 [63 to 78] | 59 [51 to 67]
  A/H3N2: Day 1: HI titers ≥1:110 | 40 [33 to 49] | 37 [29 to 45] | 43 [34 to 51] | 47 [39 to 55]
  A/H3N2: Day 50: HI titers ≥1:110 | 88 [82 to 93] | 86 [80 to 91] | 82 [74 to 88] | 97 [93 to 99]
  B: Day 1: HI titers ≥1:110 | 1 [0.016 to 4] | 0 [0 to 2] | 0 [0 to 3] | 0 [0 to 3]
  B: Day 50: HI titers ≥1:110 | 40 [33 to 49] | 30 [23 to 38] | 24 [17 to 32] | 39 [31 to 47]
  A/H1N1: Day 1: HI titers ≥1:151 | 25 [18 to 33] | 30 [23 to 38] | 26 [19 to 34] | 25 [18 to 33]
  A/H1N1: Day 50: HI titers ≥1:151 | 76 [69 to 83] | 76 [68 to 83] | 70 [62 to 78] | 58 [49 to 66]
  A/H3N2: Day 1: HI titers ≥1:151 | 40 [33 to 49] | 37 [29 to 45] | 43 [34 to 51] | 47 [39 to 55]
  A/H3N2: Day 50: HI titers ≥1:150 | 88 [82 to 93] | 86 [80 to 91] | 81 [73 to 87] | 97 [93 to 99]
  B: Day 1: HI titers ≥1:151 | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 3] | 0 [0 to 3]
  B: Day 50: HI titers ≥1:151 | 40 [32 to 48] | 30 [23 to 38] | 23 [17 to 31] | 39 [31 to 47]
  A/H1N1: Day 1: HI titers ≥1:330 | 12 [7 to 18] | 14 [9 to 21] | 11 [7 to 18] | 11 [6 to 17]
  A/H1N1: Day 50: HI titers ≥1:330 | 51 [43 to 59] | 50 [42 to 59] | 43 [35 to 52] | 34 [26 to 42]
  A/H3N2: Day 1: HI titers ≥1:330 | 16 [11 to 23] | 12 [7 to 18] | 13 [8 to 19] | 21 [15 to 29]
  A/H3N2: Day 50: HI titers ≥1:330 | 62 [53 to 69] | 56 [48 to 65] | 52 [43 to 60] | 68 [59 to 75]
  B: Day 1: HI titers ≥1:330 | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 3] | 0 [0 to 3]
  B: Day 50: HI titers ≥1:330 | 4 [2 to 9] | 4 [2 to 9] | 3 [1 to 7] | 8 [4 to 13]
  A/H1N1: Day 1: HI titers ≥1:629 | 9 [5 to 15] | 12 [7 to 18] | 11 [6 to 17] | 8 [4 to 14]
  A/H1N1: Day 50: HI titers ≥1:629 | 48 [40 to 56] | 47 [39 to 55] | 43 [35 to 52] | 33 [26 to 41]
  A/H3N2: Day 1: HI titers ≥1:629 | 16 [11 to 23] | 12 [7 to 18] | 12 [7 to 19] | 21 [15 to 29]
  A/H3N2: Day 50: HI titers ≥1:629 | 62 [53 to 69] | 56 [47 to 64] | 52 [43 to 60] | 68 [59 to 75]
  B: Day 1: HI titers ≥1:629 | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 3] | 0 [0 to 3]
  B: Day 50: HI titers ≥1:629 | 4 [2 to 9] | 3 [1 to 8] | 3 [1 to 7] | 7 [3 to 12]

9. Secondary Outcome: Percentages of Subjects (6 to <48 Months Old) Achieving MN Titer ≥1:20 After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of number (%) of subjects (6 to <48 months old) achieving MN titer ≥1:20 as measured by MN assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
  Post-vaccination MN titer ≥1:20 was defined as for subjects with baseline (day 1) MN titer <1:10, or a minimum 2-fold increase in titer on day 50 for subjects with baseline titer ≥1:10 and corresponding 95% CI
Time Frame: Day 1 and Day 50 post vaccination
Population: Analysis was done on PPS
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 156 | 148 | 141 | 147
Percentage of subjects
  A/H1N1 | 94 [89 to 97] | 93 [88 to 97] | 91 [86 to 96] | 97 [93 to 99]
  A/H3N2 | 95 [90 to 98] | 94 [89 to 97] | 94 [89 to 98] | 94 [89 to 97]
  B | 92 [86 to 95] | 92 [86 to 96] | 93 [87 to 97] | 97 [93 to 99]

10. Secondary Outcome: Percentages of Subjects (6 to <48 Months Old) Achieving MN Titer ≥1:40 After Receiving Two Doses of Either TIVc or TIVe Vaccine
Description: Immunogenicity was assessed in terms of number (%) of subjects (6 to <48 months old) achieving MN titer ≥1:40 as measured by MN assay, day 50 after vaccination with two doses of either TIVc or TIVe vaccine
  Post-vaccination MN titer ≥1:40 was defined as for subjects with baseline (day 1) MN titer <1:10, or a minimum 4-fold increase in titer on day 50 for subjects with baseline titer ≥1:10 and corresponding 95% CI
Time Frame: Day 1 and Day 50 post vaccination
Population: Analysis was done on PPS
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 156 | 148 | 141 | 147
Percentages of subjects
  A/H1N1 | 87 [80 to 91] | 89 [82 to 93] | 84 [77 to 90] | 95 [90 to 98]
  A/H3N2 | 85 [79 to 90] | 85 [78 to 90] | 82 [74 to 88] | 80 [73 to 86]
  B | 83 [76 to 88] | 87 [81 to 92] | 83 [76 to 89] | 96 [91 to 98]

11. Secondary Outcome: Number of Subjects (6 to <48 Months Old) Reporting Solicited Local (Grading Type I) and Systemic Adverse Events (AEs) After Two Doses of Either TIVc or TIVe Vaccine
Description: Safety was assessed in terms of number of subjects (6 to <48 months old) reporting solicited local and systemic reactions, day 1 to day 7 after vaccination with two doses of either TIVc or TIVe vaccine (By Any Vaccination)
Time Frame: Day 1 to Day 7
Population: Analyses was done on solicited safety data set. 4 subjects (3 subjects from the TIVe group, and 1 subject from the full dose TIVc group, were excluded from the solicited safety set analyses (6h -day3, day4-day7 and 6h - day 7) as these subjects did not provide any post vaccination solicited safety data
Measure: Number; unit: Subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 174 | 165 | 167 | 161
Subjects
  Any local AEs | 64 | 56 | 60 | 54
  Injection site tenderness | 50 | 43 | 42 | 45
  Injection site erythema | 19 | 24 | 24 | 17
  Injection site induration | 13 | 14 | 9 | 8
  Injection site ecchymosis | 9 | 9 | 7 | 7
  Any Systemic | 78 | 72 | 69 | 66
  Chills | 7 | 5 | 7 | 9
  Change in eating habits | 29 | 35 | 28 | 29
  Sleepiness | 30 | 28 | 21 | 24
  Irritability | 30 | 31 | 29 | 27
  Vomiting | 21 | 20 | 22 | 14
  Diarrhea | 31 | 31 | 29 | 34
  Fever (≥ 38°C ) | 15 | 20 | 21 | 21
  Prophylactic use of antipyretics/analgesics | 9 | 21 | 25 | 13
  Therapeutic use of antipyretics/analgesics | 17 | 21 | 24 | 22

12. Secondary Outcome: Number of Subjects (6 to <48 Months Old) Reporting Unsolicited Adverse Events (AEs) After Two Doses of Either TIVc or TIVe Vaccine
Description: Safety was assessed in terms of number of subjects (6 to <48 months old) reporting unsolicited reactions after Each /any Vaccination from Day 1 [Post Vaccination] to Day 29 [Pre Clinic Visit] and Day 29 [Post Vaccination] to Day 50 [Pre Clinic Visit] , Serious Adverse Events (SAEs), AEs leading to New Onset of Chronic Diseases (NOCD), AEs leading to withdrawal from the study and concomitant medications (day 1 to day 209) after vaccination with two doses of either TIVc or TIVe vaccine (By Any Vaccination)
Time Frame: Unsolicited AEs after Each/any Vaccination from Day 1 to Day 29 and Day 29 to Day 50 , Day 1 to Day 209
Population: Analyses was done on unsolicited safety data set i.e. all subjects in the exposed set who have post-vaccination unsolicited AE data
Measure: Number; unit: Subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe
Number analyzed (Participants) | 174 | 166 | 167 | 164
Subjects
  Any AEs(after any vaccination) | 102 | 107 | 91 | 94
  Possibly/probably related AEs (after any vaccin.) | 38 | 43 | 43 | 35
  Any AEs(after vaccination 1) | 79 | 84 | 69 | 76
  Any AEs(after vaccination 2) | 56 | 64 | 50 | 48
  Possibly/probably related AEs (after vaccination 1 | 30 | 33 | 31 | 31
  Possibly/probably related AEs (after vaccination 2 | 11 | 20 | 18 | 14
  Any SAE | 4 | 8 | 10 | 6
  Any possibly/probably related SAE | 0 | 0 | 0 | 0
  Any AE leading to premature withdrawal from study | 0 | 0 | 0 | 0
  New onset of chronic disease | 0 | 1 | 1 | 1
  Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period, up to day 209 post vaccination.
Description: Solicited AEs were collected from day 1 to day 7 post vaccination, unsolicited AEs were collected from day 1 to day 50 post vaccination and SAEs -collected from day 1 to day 209 post vaccination.
  A systematic adverse event is equivalent to an event that was solicited by the diary card, whereas a non-systematic event is an unsolicited adverse event
Groups:
- Total: Total number of subjects
Arm/Group | TIVc-High Dose | TIVc-Full Dose | TIVc- Half Dose | TIVe | Total
Serious Adverse Events (participants affected / at risk) | 4/174 | 8/166 | 10/167 | 6/164 | 28/671
Other Adverse Events (participants affected / at risk) | 142/174 | 133/166 | 141/167 | 127/164 | 543/671
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc-High Dose (N=174) | TIVc-Full Dose (N=166) | TIVc- Half Dose (N=167) | TIVe (N=164) | Total (N=671)
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 2 | 0 | 1 | 3
PHARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 2 | 2 | 0 | 4
VARICELLA (Infections and infestations) | 0 | 0 | 0 | 1 | 1
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1 | 5
FEBRILE CONVULSION (Nervous system disorders) | 1 | 2 | 1 | 3 | 7
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 3
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
AMOEBIASIS (Infections and infestations) | 0 | 0 | 1 | 1 | 2
GASTROENTERITIS (Infections and infestations) | 2 | 0 | 1 | 1 | 4
HAND-FOOT-AND-MOUTH DISEASE (Infections and infestations) | 0 | 0 | 0 | 1 | 1
PERIORBITAL CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc-High Dose (N=174) | TIVc-Full Dose (N=166) | TIVc- Half Dose (N=167) | TIVe (N=164) | Total (N=671)
DIARRHOEA (Gastrointestinal disorders) | 32 | 32 | 30 | 36 | 130
VOMITING (Gastrointestinal disorders) | 21 | 20 | 22 | 14 | 77
INFLUENZA LIKE ILLNESS (General disorders) | 20 | 38 | 35 | 37 | 130
INJECTION SITE ERYTHEMA (General disorders) | 30 | 36 | 32 | 29 | 127
INJECTION SITE HAEMORRHAGE (General disorders) | 9 | 10 | 8 | 7 | 34
INJECTION SITE INDURATION (General disorders) | 13 | 16 | 12 | 10 | 51
INJECTION SITE PAIN (General disorders) | 56 | 48 | 47 | 47 | 198
PYREXIA (General disorders) | 22 | 28 | 32 | 22 | 104
NASOPHARYNGITIS (Infections and infestations) | 19 | 17 | 22 | 25 | 83
RHINITIS (Infections and infestations) | 22 | 30 | 19 | 26 | 97
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 48 | 44 | 53 | 41 | 186
SOMNOLENCE (Nervous system disorders) | 30 | 28 | 21 | 24 | 103
EATING DISORDER (Psychiatric disorders) | 29 | 35 | 28 | 29 | 121
IRRITABILITY (Psychiatric disorders) | 34 | 37 | 34 | 29 | 134
CHILLS (General disorders) | 7 | 5 | 7 | 9 | 28
BRONCHITIS (Infections and infestations) | 6 | 11 | 12 | 12 | 41
Gastroenteritis (Infections and infestations) | 17 | 17 | 15 | 15 | 64
Impetigo (Infections and infestations) | 6 | 8 | 10 | 6 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less